CLINICAL TRIAL: NCT02362451
Title: A Randomized, Placebo-Controlled Phase II Study of Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Men With Stage D0 Prostate Cancer
Brief Title: Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Men With Stage D0 Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150075; 15-C-0075
Record Dates: First submitted 2015-02-12; First posted 2015-02-13 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Dendritic Cell Vaccine; Multi Epitope Tarp Peptide; Autolougous Dendritic Cell; D0 Prostate Cancer; Vaccine Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TARP; Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment (Experimental): All patients to receive autologous multi-epitope T-cell receptor g alternate reading frame protein (TARP) DC vaccine before randomization
  Interventions: Biological: Multi-epitope (ME) T-cell receptor g alternate reading frame protein (TARP) vaccine
- 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment (Experimental): Autologous multi-epitope T-cell receptor g alternate reading frame protein (TARP) DC vaccine after randomization
  Interventions: Biological: Multi-epitope (ME) T-cell receptor g alternate reading frame protein (TARP) vaccine
- 3/Placebo (Placebo Comparator): Autologous elutriated monocyte vaccine placebo after randomization
  Interventions: Biological: Autologus elutriated monocyte placebo vaccine

INTERVENTIONS:
Biological: Autologus elutriated monocyte placebo vaccine — 20x10^6 viable cells/dose at weeks 3, 6, 9, 12, 15 and 24
  Arms: 3/Placebo
Biological: Multi-epitope (ME) T-cell receptor g alternate reading frame protein (TARP) vaccine — 20x10^6 viable cells/dose at weeks 3, 6, 9, 12, 15 and 24
  Arms: 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment; 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment

SUMMARY:
Background:

- Men who continue to have an elevated or rising prostate specific antigen (PSA) level after their primary prostate cancer treatment are at increased risk for their cancer to progress. The time it takes to progress is highly variable. One way to predict this progression is based on the change in PSA levels over time. This is called the PSA doubling time (PSADT). Researchers want to test a vaccine on men with Stage D0 prostate cancer. Stage D0 means the PSA has become detectable again or has started to rise after primary treatment, but has not spread to other organs.

Objectives:

- To test a vaccines effectiveness on the rate of PSA increase using PSADT and tumor growth rates.

Eligibility:

- Men with Stage D0 prostate cancer with a PSADT between 3 and 15 months.

Design:

* Participants will be screened with blood tests, scans, physical exam, and medical history. Their prostate cancer will be confirmed.
* Participants will undergo apheresis. Blood will be removed with a needle from one arm. A machine will separate the white blood cells. The blood, minus the white cells, will be returned through a needle in the other arm.
* Participants will have 14 visits. At each visit, they will have a physical exam and blood tests. They will discuss any side effects.
* Participants will get injections of either the vaccine or placebo at weeks 3, 6, 9, 12, 15, and 24. Both will be made from the participants own cells.
* Participants will be selected randomly to receive either active vaccine or placebo. For every two participants assigned to active vaccine, one participant will be assigned to placebo vaccine.
* Participants will get a Vaccine Report Card to to complete after receiving vaccine.
* The study lasts 96 weeks.

DETAILED DESCRIPTION:
TARP

* T-cell receptor g alternate reading frame protein (TARP) is a 58 amino acid protein expressed by both normal and malignant prostate cancer tissue; 95% of prostate cancer specimens are positive for TARP expression. TARP is highly expressed in prostate cancers of all Gleason types, in primary as well as metastatic disease, and in hormone sensitive and castrate resistant prostate cancer. Therefore, TARP is an ideal tumor antigen target for a vaccine.
* A prospective, randomized pilot study of 1st generation TARP Peptide vaccination (National Cancer Institute (NCI) 09-C-0139) utilizing TARP WT 27-35 and EE29-37-9V peptides was conducted in human leukocyte antigen serotype within the HLA-A serotype group (HLA-A 0201) positive men with stage D0 prostate cancer (prostate specific antigen (PSA) biochemical recurrence) and a PSA doubling time (PSADT) of greater than or equal to 3 months and less than or equal to 15 months. TARP vaccination was found to be immunogenic, safe and well tolerated, with adverse events limited to injection site reactions less than or equal to Grade 2. TARP vaccination was also associated with a decreased slope log PSA compared to pre-vaccination baseline in 72% of subjects reaching 24 weeks and 74% reaching 48 weeks (p=0.0012 and p=0.0004 for overall changes in slope log PSA, respectively); TARP vaccination also resulted in a 50% decrease in calculated tumor growth rate constant: pre-vaccine g = 0.0042/day, post-vaccine g = 0.0021/day (p=0.003); TARP-specific interferon gamma (IFN-g) enzyme-linked immune absorbent spot (ELISPOT) responses were detected in the majority of subjects but did not correlate with decreases in slope log (PSA).

Multi-Epitope (ME) TARP Vaccine

* The vaccine platform includes the original two 9-mer HLA-A*0201 binding TARP peptide epitopes (WT27-35 and EE29-37-9V) utilized in NCI 09-C-0139 as well as an additional five 20-mer TARP peptides overlapping by 10 amino acids for a total of 7 peptides that span the amino acid sequence of the entire TARP protein.
* The advantage of this multi-epitope TARP peptide vaccine platform is that the overlapping epitopes cover the entire TARP protein, resulting in potential for induction of a multi-valent anti-TARP response. In addition, these longer synthetic peptides include TARP-specific major histocompatibility complex (MHC)class II cluster of differentiation 4 (CD4)+ T cell helper epitopes that will allow generation of better cluster of differentiation 8 (CD8)+ T cell responses with improved functional avidity and longevity as well as humoral anti-TARP antibody responses.

Study Objectives:

Primary:

-To assess the difference in the slope log (PSA) for Weeks3-24 minus that formed for the 12 months prior to enrollment on study (referred to as slope324 pre-slope) as well as the slope log (PSA) for weeks 3-48 versus the same pre-treatment slope log (PSA) (referred to as slope 348 preslope) in patients na(SqrRoot) ve to TARP vaccination receiving active, multi-epitope TARP vaccination vs. placebo.

Eligibility:

* Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate.
* Stage D0 disease with documented biochemical progression documented by rising PSA and no evidence of metastatic disease by physical examination, computed tomography (CT) scan or bone scan.
* Prostate specific antigen doubling time (PSADT) greater than or equal to 3 months and less than or equal to 15 months:

  ----Patients must have greater than or equal to 3 PSA measurements over greater than or equal to 3 months.

  --- The interval between PSA measurements must be greater than or equal to 4 weeks.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1.
* No other concurrent anticancer therapy or prior prostate cancer vaccines expressing TARP.

Study Design:

* Phase II, prospective, single-blinded, randomized, placebo controlled study of 96 weeks duration in men with Stage D0 prostate cancer. Men with a PSADT greater than or equal to 3 months and less than or equal to 15 months will be randomized 2:1 to receive multi-epitope (ME) TARP autologous dendritic cell (DC) vaccination or a control eleutriated monocyte vaccine placebo.
* An initial lead-in of 6 patientswill be enrolled to allow preliminary assessment of the safety of the ME TARP vaccine platform through 12 weeks before enrollment of prospectively randomized subjects blinded to treatment assignment begins.
* All patients will receive a total of 6 doses of vaccine (20 x10(6) viable cells/dose) delivered intradermally at Weeks 3, 6, 9, 12, 15, and 24. All patients will undergo a 15-18L apheresis at Week 0 and restaging at Weeks 48 and 96 to confirm maintenance of Stage D0 disease.

Sample size: N = 72 (6 lead-in patients for safety assessment, 2:1 randomization: TARP N = 44; placebo N =22).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate. Histology confirmation must be documented with a formal pathology report. Notes from an outside physician describing the pathologic findings (based on a prior review of the full pathology report) may be used if unable to obtain the original pathology report. This will eliminate the need for an additional invasive tissue biopsy.
2. Must have completed and recovered from all prior definitive therapy (surgery, brachytherapy, cryotherapy or radiotherapy) for the primary tumor, or other definitiveintent local therapy.
3. Stage D0 disease with documented biochemical progression documented by rising prostate specific-antigen (PSA) and no evidence of metastatic disease by physical examination, computed tomography (CT) scan or bone scan.
4. Prostate specific-antigen doubling time (PSADT) greater than or equal to 3 months and less than or equal to 15 months:

   * Patients must have greater than or equal to 3 PSA measurements over greater than or equal to 3 months.
   * The interval between PSA measurements must be greater than or equal to 4 weeks.
5. For patients following definitive radiation therapy or cryotherapy: a rise in PSA of > 2ng/mL above the nadir (per Radiation Therapy Oncology Group (RTOG)-American Society for Therapeutic Radiology and Oncology (ASTRO) consensus criteria).
6. For patients following radical prostatectomy: 2 absolute PSA values > 0.2ng/ml.
7. Non-castrate level of testosterone: greater than or equal to 50 ng/dL (prior antiandrogen treatment (ADT) allowed; must be greater than or equal to 6 months since last dose of ADT).
8. Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1.
9. Hemoglobin greater than or equal to 9.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500/mm(3), absolute lymphocyte count (ALC) greater than or equal to 500/ mm(3), absolute neutrophil count (ANC) greater than or equal to 1,000/mm(3) platelet count greater than or equal to 75,000/mm(3), and prothrombin time (PT)/Partial thromboplastin time (PTT)PTT less than or equal to 1.5 times upper limit of normal (ULN) unless receiving clinically indicated anticoagulant therapy; serum glutamic-pyruvic transaminase (SGPT)/Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 3 times ULN, total bilirubin less than or equal to 1.5 times ULN; creatinine less than or equal to 1.5 times ULN and estimated GFR (eGFR) greater than or equal to 60 ml/min.
10. Hepatitis B and C negative (unless the result is consistent with prior vaccination or prior infection with full recovery); human immunodeficiency virus (HIV) negative.
11. No use of investigational agents within 4 weeks of study enrollment or use of immunosuppressive or immunomodulating agents within 8 weeks of study entry.
12. No other concurrent anticancer therapy or prior prostate cancer vaccines expressing T-cell receptor alternate reading frame protein (TARP).
13. No alternative medications or nutriceuticals known to alter PSA (e.g. phytoestrogens and saw palmetto). Note: patients receiving medications for urinary symptoms such as Flomax or 5-alpha reductase inhibitors (finasteride and dutasteride) on a chronic stable dose for at least 3 months prior to study enrollment are allowed.

EXCLUSION CRITERIA:

1. Patients with an active second malignancy other than adequately treated squamous or basal cell carcinoma of the skin.
2. Patients with active infection.
3. Patients on immunosuppressive therapy including:

   - Systemic corticosteroid therapy for any reason. Patients receiving inhaled or topical corticosteroids may participate.
4. Other significant or uncontrolled medical illness. Patients with a remote history of asthma or active mild asthma may participate.
5. Patients who, in the opinion of the Principal Investigator, have significant medical or psychosocial problems that warrant exclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All collected individual participant data (IPD) will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0075.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled to the Arm 3 placebo group.
Groups:
- 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment: Cohort 1 All patients to receive autologous multi-epitope T-cell receptor g alternate reading frame protein (TARP) DC vaccine before randomization
  Multi-epitope (ME) T-cell receptor g alternate reading frame protein (TARP) vaccine: 20x10^6 viable cells/dose at weeks 3, 6, 9, 12, 15 and 24
- 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment: Cohort 2 Autologous multi-epitope T-cell receptor g alternate reading frame protein (TARP) DC vaccine after randomization
  Multi-epitope (ME) T-cell receptor g alternate reading frame protein (TARP) vaccine: 20x10^6 viable cells/dose at weeks 3, 6, 9, 12, 15 and 24
Period: Overall Study
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment
Started | 6 | 1
Completed | 2 | 0
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Progression | 1 | 0
Not completed — Participant chose other therapy. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.73 (3.5) | 57.2 (0) | 67.09 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in the Slope Log of Prostate-specific Antigen Pre vs Post Treatment
Description: PSA Doubling Time (PSADT) and slope log (PSA) were calculated at every study visit using the PSADT Memorial Sloane Kettering nomogram. The values were calculated to demonstrate the rate of rise of PSA, expressed as the velocity in nanograms/mL/year, or the PSA doubling time, in months or years. PSA is a tumor marker for prostate cancer and after surgery (undetectable - e.g. <0.2 ng/mL) or radiation PSA should fall to a very low level when the disease is effectively treated. When PSA increases (>2.0 ng/mL) after surgery or radiation that could mean recurrence of the disease. If prostate cancer is growing slower or shrinking after the treatment, PSADT can be longer while PSA slope log is shorter as tumor will make less PSA.
Time Frame: One year pre-enrollment; weeks 3-24, and 3 - 48 post vaccine
Population: One participant in the lead in group had no data for week 48 due to other treatment, thus data could not be used. And one participant in the active group had no data for week 3-24 and 3-48 due to other treatment, thus data could not be used.
Measure: Median (Full Range); unit: slope log
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment
Number analyzed (Participants) | 6 | 1
slope log
  Pre treatment | 0.07 [0.05 to 0.19] | 0.05 [0 to 0.05]
  Weeks 3-24: number analyzed (Participants) | 6 | 0
  Weeks 3-24 | 0.08 [-0.01 to 0.21] |
  Weeks 3-48: number analyzed (Participants) | 5 | 0
  Weeks 3-48 | 0.06 [0.01 to 0.07] |

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of vaccine treatment to time of progression or death. Given the study population in biochemically recurrent prostate cancer, progression is defined as 1)"radiographic progression" by computed tomography (CT) or bone scan, 2) prostate-specific antigen doubling time (PSADT) that is 3 month or shorter, 3) PSADT decrease 50% or more compared to enrollment PSADT.
Time Frame: Week 96 after initial vaccination
Measure: Median (Full Range); unit: Weeks
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment
Number analyzed (Participants) | 6 | 1
Weeks | 96 [48 to 96] | NA [NA to NA] — The median and full range is not available for the 1 participant in the Active group. The participant was censored at that time point because he came off study, not that he progressed.]

3. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 54 months and 13 days for cohort 1 and 5 months and 9 days for cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment
Number analyzed (Participants) | 6 | 1
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 54 months and 13 days for cohort 1 and 5 months and 9 days for cohort 2.
Arm/Group | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Lead-in T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment (N=6) | 2/Active T-cell Receptor g Alternate Reading Frame Protein Dendritic Cell (DC) Vaccine Treatment (N=1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chills (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 6 (71) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle aches/ left thigh (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Discoloration. Left and right forearm at the injection sites.
Skin and subcutaneous tissue disorders - Other, lesion on scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, small nodule behind right ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — wo hyperkeratotic lesions on left arm at the injection site.
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT02362451/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Affected Patient (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT02362451/ICF_001.pdf
  • Informed Consent Form: Addendum 1 to 15C0075 (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02362451/ICF_002.pdf
  • Informed Consent Form: Addendum 2 to 15C0075 (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT02362451/ICF_003.pdf